CLINICAL TRIAL: NCT00802100
Title: Comparison of Optimal Antipsychotic Treatments for Schizophrenia Pilot Study
Brief Title: Comparison of Optimal Antipsychotic Treatments for Adults With Schizophrenia
Acronym: COATS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N01 MH090001-02; N01MH90001 (NIH); N01MH090001 (NIH)
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2012-04

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Perphenazine; Aripiprazole; Metformin; Simvastatin; Benztropine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Olanzapine (Experimental): Participants will receive treatment with olanzapine and metformin, with the possible addition of simvastatin or benztropine, depending on side effects.
  Interventions: Drug: Olanzapine; Drug: Metformin; Drug: Simvastatin; Drug: Benztropine
- Perphenazine (Experimental): Participants will receive treatment with perphenazine and benztropine, with the possible addition of simvastatin or metformin, depending on side effects.
  Interventions: Drug: Perphenazine; Drug: Metformin; Drug: Simvastatin; Drug: Benztropine
- Aripiprazole (Experimental): Participants will receive treatment with aripiprazole, with the possible addition of simvastatin, metformin, or benztropine, depending on side effects.
  Interventions: Drug: Aripiprazole; Drug: Metformin; Drug: Simvastatin; Drug: Benztropine

INTERVENTIONS:
Drug: Olanzapine — Daily tablets of 10 to 30 mg
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Perphenazine — Daily tablets of 8 to 24 mg
  Other Names: Trilafon
  Arms: Perphenazine
Drug: Aripiprazole — Daily tablets of 10 to 30 mg
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Metformin — Daily tablets of 850 to 2550 mg
  Other Names: Glucophage
Drug: Simvastatin — Daily tablets of 20 to 40 mg
  Other Names: Zocor
Drug: Benztropine — Daily tablets of 1 to 2 mg
  Other Names: Cogentin

SUMMARY:
This study will compare the safety and effectiveness of three different antipsychotic medications, as well as the use of other medications to limit treatment side effects, in adults with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic brain disease affecting approximately 1% of Americans. Antipsychotic medications can treat some of the most severe symptoms of schizophrenia, but they are not a cure, are often taken for long periods of time, and can have severe side effects. Other, secondary medications can provide relief from some of the most common severe side effects. This study will compare the safety and effectiveness of three different antipsychotic medications, as well as the use of additional medications to limit treatment side effects, in adults with schizophrenia.

Participation in this study will last 28 to 30 weeks and include 11 visits to a study clinic. Each visit will last 2 to 3 hours. The first 2 visits will include screening and baseline measurements. The screening visit will take place at study entry, and the baseline visit will take place 3 to 14 days later. Study visits will then occur 1, 2, and 4 weeks after the baseline visit, followed by monthly visits.

At the baseline visit participants will be randomly assigned to receive olanzapine, perphenazine, or aripiprazole for 28 weeks. Dosage for all three antipsychotic medications will start at low levels and be increased to full strength over 2 weeks. If participants are taking another antipsychotic when they enter the study, this 2-week period will also be used to slowly reduce and then end treatment with the non-study antipsychotic. Side effects to all three antipsychotics will be monitored, and, depending on the side effect, one of three different medications will be added to the treatment regimen. If increased cholesterol levels are experienced with any antipsychotic, simvastatin will be added; if weight gain is experienced, metformin will be added; if involuntary movements, inner restlessness, or muscle stiffness are experienced, benztropine will be added. Because of already known side effects, participants assigned to olanzapine or perphenazine will automatically add metformin or benztropine, respectively, to their regimens.

Starting on the third study visit, participants will also undergo a behavioral treatment aimed at reducing cardiovascular risk factors. This behavioral treatment will involve nine 20-minute sessions, with phone calls being made to participants between sessions.

During each study visit, assessments will be made of schizophrenia symptoms, side effects, adherence to medication regimen, vital signs, waist circumference, and weight. Participants will also complete a questionnaire on use of health care services and undergo instructions on exercise and eating right. On visits 1, 5, 7, and 11, blood will be drawn for standard lab tests. Additional measures at the screening visit will include questions about medical and psychiatric history, a urine test for drugs, and a questionnaire about physical and social activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder, as defined by DSM-IV-TR criteria and confirmed by the Structured Clinical Interview for DSM-IV (SCID)
* Treated with antipsychotic medication for less than 5 years
* Adequate decisional capacity to make a choice about participating in this research study. Adequate decisional capacity will be determined through the aid of a 10-item decisional capacity quiz adapted from the University of California, San Diego, Brief Assessment of Capacity to Consent (UBACC) scale.
* Psychotic exacerbation within the month prior to study entry that required psychiatric hospitalization or an increased level of care
* Willing to use an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study. Acceptable methods include oral, injectable, or implanted contraceptives; intrauterine devices; or barrier methods, such as condoms, diaphragm, and spermicides.

Exclusion Criteria:

* Body mass index at or above 35 kg/m2 or below 18 kg/m2
* Hemoglobin A1c level at or above 7%
* Hematocrit level at or above 31%
* Non-high density lipoprotein cholesterol at or above 190 mg/dL
* Triglycerides at or above 500 mg/dL
* Documented failure, defined as inefficacy or intolerability, with an adequate trial of olanzapine, perphenazine, or aripiprazole. Adequate trials last at least 4 weeks at a minimum dose of 15 mg/day of aripiprazole, 15 mg/day of olanzapine, or 16 mg/day of perphenazine.
* Current treatment with olanzapine, perphenazine, or aripiprazole for more than 1 month
* Known hypersensitivity to metformin, simvastatin, or benztropine
* Treatment with a medication prescribed for weight loss
* Diagnosis of diabetes mellitus or treatment with insulin or other diabetes medication
* Contraindications to metformin use, including any of the following:

  * Diagnosis of congestive heart failure
  * Renal impairment, defined as serum creatinine at or above 1.5 in males and 1.4 in females, or creatinine estimated glomerular filtration rate (GFR) outside of normal limits
  * Hepatic disease, defined as aspartate transaminase (AST), alanine transaminase (ALT), or c-glutamyl transferase (CGT) more than 1.5 times upper limit of normal (ULN) or total bilirubin more than 1.2 times ULN
  * Metabolic acidosis, defined as a serum CO2 level less than the lower limit of normal
  * Recent (in the past 30 days) or scheduled radiological studies involving iodinated contrast material
  * Alcohol abuse or dependence, as determined by SCID within the past month
  * Concurrent treatment with certain drugs known to increase metformin blood levels
* Any unstable or serious medical condition, as judged by the investigator
* Pregnant or breastfeeding
* Diagnosis of mental retardation or delirium, as defined by the DSM-IV-TR

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Swartz, MD, Principal Investigator — Duke University; T. Scott Stroup, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Joseph P. McEvoy, MD, Principal Investigator — Duke University
Locations (13):
- United States (13):
  - SHANTI Clinical Trials, Colton, California
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Clinical Insights, Glen Burnie, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of Minnesota School of Medicine, Minneapolis, Minnesota
  - Research Foundation for Mental Hygiene, New York, New York
  - Duke University Medical Center-John Umstead Hospital, Butner, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This feasibility-focused pilot study was conducted at 14 clinical sites affiliated with the Schizophrenia Trials Network in 2008-9.
Groups:
- Olanzapine: Participants will receive treatment with olanzapine and metformin, with the possible addition of simvastatin or benztropine, depending on side effects.
  Olanzapine dose 10-30 mg/day Metformin dose 850-2550 mg/day
- Perphenazine: Participants will receive treatment with perphenazine and benztropine, with the possible addition of simvastatin or metformin, depending on side effects.
  Perphenazine dose 8-24 mg/day Benztropine dose 1-2 mg/day Metformin dose 850-2550 mg/day Simvistatin dose 20-40 mg/day
- Aripiprazole: Participants will receive treatment with aripiprazole, with the possible addition of simvastatin, metformin, or benztropine, depending on side effects.
  Aripiprazole dose 10-30 mg/day Benztropine dose 1-2 mg/day Metformin dose 850-2550 mg/day Simvistatin dose 20-40 mg/day
Period: Overall Study
Arm/Group | Olanzapine | Perphenazine | Aripiprazole
Started | 6 | 9 | 6
Completed | 0 | 2 | 2
Not Completed | 6 | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Perphenazine | Aripiprazole | Total
Number analyzed (Participants) | 6 | 9 | 6 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 30 (9.7) | 30 (8.1) | 27 (7.9) | 29 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 8
  Male | 4 | 5 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Randomizing a Cohort of Participants Meeting the Inclusion and Exclusion Criteria of the Study
Description: Goal was to randomize 60 participants who met eligibility criteria.
Time Frame: Baseline
Population: Total study population
Measure: Number; unit: participants
Groups:
- Overall Study: This refers to the feasibility of the entire pilot study. Only 21 eligible participants of the goal of 60 were randomized because sites were unable to identify adequate numbers of eligible participants.
Arm/Group | Overall Study
Number analyzed (Participants) | 21
participants | 21

2. Secondary Outcome: Antipsychotic Efficacy, Defined as Completion of the Trial Without Psychiatric Hospitalization, Clinician Decision to Discontinue Treatment, or Patient Decision to Discontinue Treatment
Time Frame: Measured over 28 weeks of study visits
Population: Analysis population is those randomized. Outcome is discontinuation from study treatment before 28 weeks
Measure: Number; unit: participants
Arm/Group | Olanzapine | Perphenazine | Aripiprazole
Number analyzed (Participants) | 6 | 9 | 6
participants
  Inefficacy | 0 | 1 | 1
  Unacceptable side effects | 0 | 0 | 0
  Patient refusal | 3 | 0 | 0
  Drop-out, no information available | 2 | 1 | 0
  Administrative | 1 | 5 | 3
  Completed trial without discontinuing | 0 | 2 | 2

ADVERSE EVENTS:
Arm/Group | Olanzapine | Perphenazine | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/9 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=6) | Perphenazine (N=9) | Aripiprazole (N=6)
Exacerbation of Schizophrenia (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Uterine fibroids (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine (N=6) | Perphenazine (N=9) | Aripiprazole (N=6)
Akathisia/activation (Psychiatric disorders) | 4 (4) | 7 (7) | 6 (6)
Sleepiness (General disorders) | 3 (3) | 9 (9) | 5 (5)
Weight gain (General disorders) | 3 (3) | 8 (8) | 6 (6)
Dry mouth (General disorders) | 3 (3) | 6 (6) | 5 (5)
Increased appetite (General disorders) | 1 (1) | 6 (6) | 6 (6)
Insomnia (General disorders) | 2 (2) | 7 (7) | 4 (4)
Akinesia (General disorders) | 2 (2) | 5 (5) | 5 (5)
Hypersomnia (General disorders) | 2 (2) | 4 (4) | 4 (4)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4)
Orthostatic faintness (Cardiac disorders) | 1 (1) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Decreased sex drive (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 4 (4)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Diminished sexual arousal (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 3 (3)
sialorrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Urinary hesitancy (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Gynecomastia/galactorrhea/ (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 2 (2)
Menstrual irregularities (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 2 (2)
Problem with sexual orgasm (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 2 (2)
Incontinence/nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
It was determined in this pilot study that the existing procedures and eligibility criteria could not be adequately implemented and that a larger-scale study was not feasible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No